CLINICAL TRIAL: NCT06916234
Title: Evaluation of the Analgesic Efficacy of the Combination of Dexketoprofen + Paracetamol and the Combination of Naproxen Sodium + Codeine in Patients With Acute Dental Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ibrahim doğru (Other)
Responsible Party: Sponsor-Investigator, ibrahim doğru, assistant professor, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 30.11.2022/07
Record Dates: First submitted 2025-03-21; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Acute Dental Pain
MeSH Terms: interventions — dexketoprofen trometamol; Acetaminophen; Naproxen; Codeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexketoprofen Trometamol + Paracetamol (25mg + 300mg, 2x1) (Active Comparator)
  Interventions: Drug: Dexketoprofen Trometamol + Paracetamol
- Naproxen Sodium + Codeine Phosphate (550 mg + 30 mg, 2X1) (Active Comparator)
  Interventions: Drug: Naproxen Sodium + Codeine Phosphate

INTERVENTIONS:
Drug: Dexketoprofen Trometamol + Paracetamol — Dexketoprofen Trometamol + Paracetamol (25mg + 300mg) is a NSAID. It was given to the patients twice a day.
  Arms: Dexketoprofen Trometamol + Paracetamol (25mg + 300mg, 2x1)
Drug: Naproxen Sodium + Codeine Phosphate — Naproxen Sodium + Codeine Phosphate (550mg + 30mg) is a NSAID. It was given to the patients twice a day.
  Arms: Naproxen Sodium + Codeine Phosphate (550 mg + 30 mg, 2X1)

SUMMARY:
Acute dental pain is one of the most challenging conditions to treat and manage in dental practice. The aim of this study was to compare the efficacy of naproxen sodium + codeine phosphate (550/30 mg) and dexketoprofen trometamol + paracetamol (25/300 mg) in the treatment of acute dental pain in individuals with acute pericoronitis caused by impacted wisdom teeth.

DETAILED DESCRIPTION:
This randomised, prospective, single-blind study was conducted on patients who presented to Van Yuzuncu Yil University Faculty of Dentistry, Department of Oral and Maxillofacial Surgery between January 2023 and December 2023 with the complaint of acute pericoronitis originating from the lower impacted third molar teeth. At the first visit, the patients underwent a clinical examination to evaluated the patients' complaints, whether the complaints were caused by impacted lower third molar , and the presence of infection. For radiographic assessment, panoramic radiographs were taken of the region of the impacted lower third molars about which the patients complained. Patients who met the inclusion criteria were randomised into two groups, by the research assistants using the Research Randomizer (version 4.0) program to ensure blinding of the surgeons. Group A (active control group) received 550 mg naproxen sodium + 30 mg codeine phosphate and group B (research group) received 25 mg dexketoprofen trometamol + 300 mg paracetamol 2 times daily for 7 days; and amoxicillin 500 mg 3 times daily for 5 days in addition to analgesics for infection control due to acute pericoronitis. Paracetamol 500 mg was administered as rescue medication. Patients were instructed not to take rescue medication unless they had to and, if they did, to record the time and number of doses on the form given to them. Patients in the study groups received the first dose of the drugs from us and continued to receive subsequent doses every 12 hours.

A Visual Analogue Scale (VAS) with numbers ranging from 0 - no pain to 10 - un-bearable pain was used to evaluate pain. Patients were asked to record their VAS score on the form at the 6th hour (T1), 12th hour (T2), 18th hour (T3), 24th hour (T4), 2nd day (T5), 3rd day (T6), 4th day (T7), 5th day (T8), 6th day (T9) and 7th day (T10) after the first dose (T0 of study drug. Obtained data was analyzed and evaluated statistically.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 and over
2. Individuals with systemic status ASA0 and ASA1 according to the American Society of Anaesthesiologists (ASA) classification,
3. Individuals with semi-erupted impacted lower third molar teeth associated with acute pericoronitis,
4. Individuals with a VAS score of 5 and above at the first visit.

Exclusion Criteria:

1. pregnant or lactating women,
2. smokers,
3. alcohol and/or drug users,
4. those who did not attend post-operative check-ups,
5. those who were using other than the recommended medication,
6. those who developed adverse drug reactions during the study and discontinued medication,
7. those who were allergic to the study drugs,
8. those who underwent additional dental treatment during the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Pain Evaluation | 6th hour
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | 12th hour
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | 18th hour
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | 24th hour
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | 2nd day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | 3rd day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | 4th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | 5th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | 6th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | 7th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: ibrahim doğru Assist. Prof., Principal Investigator — ibrahimdogru@yyu.edu.tr
Locations (1):
- Van Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dogru I, Cigerim L. Comparison of the analgesic efficacy of dexketoprofen trometamol and paracetamol with naproxen sodium and codeine phosphate combinations in acute toothache. Sci Rep. 2025 Oct 17;15(1):36381. doi: 10.1038/s41598-025-20361-7. PMID 41107344

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT06916234/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT06916234/ICF_001.pdf